CLINICAL TRIAL: NCT01670669
Title: An Open-label Follow-up Study of 0.01 mg/kg/Day to 0.03 mg/kg/Day Prucalopride (R108512) Oral Solution in Paediatric Subjects, Aged >= 4 to <= 12 Years With Functional Faecal Retention (FFR), Who Participated in the PRU-USA-12.
Brief Title: Prucalopride in Paediatric Subjects, With Functional Faecal Retention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Movetis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRU-USA-24
Record Dates: First submitted 2012-07-31; First posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

ARMS (1):
- prucalopride (Active Comparator): 0.01 mg/kg/day to 0.03 mg/kg/day prucalopride (R108512) oral solution
  Interventions: Drug: prucalopride

INTERVENTIONS:
Drug: prucalopride — 0.01 mg/kg/day to 0.03 mg/kg/day prucalopride (R108512) oral solution

SUMMARY:
The purpose of this study is characterize the efficacy, safety, tolerability, and steady-state plasma levels after once-daily oral dosing of prucalopride (R108512) as a solution, 0.01 mg/kg to 0.03 mg/kg, given to paediatric subjects with functional faecal retention (FFR) for 8 weeks.

Hypothesis:

Pharmacokinetic profile of prucalopride in paediatric subjects is expected to resemble the adult pharmacokinetic profile. Safety and tolerability profile are expected to resemble the adult profile.

DETAILED DESCRIPTION:
This is a multicentre, open-label trial in which paediatric subjects (ages 4 to 12 years) with FFR were administered prucalopride in oral solution once daily for 8 weeks. Subjects who entered this extension trial had completed PRU-USA-12, a single-dose pharmacokinetic trial, usually within the previous week.

Evaluations for efficacy, safety and tolerability were performed, and plasma samples for analysis of prucalopride levels were obtained at 2, 4, 6 and 8 weeks.

The initial dosage of prucalopride oral solution was 0.02 mg/kg/day. Dependent on the subject's response, the parent could adjust the dosage within a range of 0.01 mg/kg/day to 0.03 mg/kg/day.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the PRU-USA-12 pharmacokinetic trial
* Subject bowels had been "cleaned-out" (ie, any faecal impactions removed)
* Written informed consent, signed by the subject's legal guardian and by the investigator
* Subject assent documented in the form of a note-to-file in the subject's source documentation

Exclusion Criteria:

• No exclusion criteria

Ages: 4 Years to 12 Years
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 1998-11; Primary Completion 1999-07 (Actual); Study Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Adverse events
  Adverse events (AEs) to be recorded by spontanous reporting or after non-leading questioning i.e. reporting of all AEs and its duration during the course of the trial. In addition at bi-weekly visits laboratory assessments, vitals signs, ECGs and physical examinations, reported as mean values and clinical significant abnormalities to be tabulated.
  Efficacy: reporting of bowel movements and its characteristics in a diary.
Efficacy
  Reporting of bowel movement frequency, i.e. average number of bowel movements on a weekly base.

SECONDARY OUTCOMES:
Secondary efficacy variables: steady-state plasma levels after once-daily oral dosing of prucalopride (R108512) as a solution, 0.01 mg/kg to 0.03 mg/kg, given to paediatric subjects with functional faecal retention (FFR) for 8 weeks. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harald Winter, M.D., Principal Investigator — Massachusetts General Hospital for Children, Boston, Massachusetts, USA

REFERENCES:
- [Derived] Winter HS, Di Lorenzo C, Benninga MA, Gilger MA, Kearns GL, Hyman PE, Vandeplassche L, Ausma J, Hoppenbrouwers M. Oral prucalopride in children with functional constipation. J Pediatr Gastroenterol Nutr. 2013 Aug;57(2):197-203. doi: 10.1097/MPG.0b013e318292f9ea. PMID 23535761